CLINICAL TRIAL: NCT02636777
Title: Predictors of Self-management in Patients With Chronic Low Back Pain
Status: Completed | Type: Observational
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Other Study IDs: 15084; 188664 (Other: IRAS Project ID)
Record Dates: First submitted 2015-12-15; First posted 2015-12-22 (Estimated); Last update posted 2018-06-21 (Actual); Status verified 2018-06

CONDITIONS: Low Back Pain
Keywords: low back pain; chronic pain; self-management; longitudinal study; predictive modelling
MeSH Terms: conditions — Low Back Pain; Chronic Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: no intervention — Patients will be allowed to continue their usual treatment as recommended by their care team.

SUMMARY:
Supported self-management (SM) is one of the key recommendations in management of chronic low back pain (CLBP). SM programmes for patients with CLBP have failed to show clinically meaningful improvement in pain and disability markers, which potentially reflect the lack of treatment matching of SM programmes. Patient selection for a SM programme for patients with CLBP is particularly difficult due to lack of extensive research on what predicts SM and its change. The overarching purpose of this study is to identify predictors of SM and its change over time in patients with CLBP. This study is a prospective non-experimental longitudinal study.

DETAILED DESCRIPTION:
Materials and methods: Patients will be recruited at baseline from the physiotherapy outpatient clinics. Three different methods have been planned to identify suitable patients in this study: from the outpatient clinics, through advertisements and therapist referrals to the study. All willing participants will be screened against the study selection criteria. Eligible participants will be provided with a pre-approved information sheet and verbal explanation about the study before obtaining written consent. The consenting patients will be requested to fill in the baseline questionnaire. The patients will be requested to fill the follow up questionnaire after six months from their baseline data collection via an online, telephone or paper-based questionnaire depending on their preference. Data required for the necessary agreement between paper-based and online or telephone survey, will be collected from up to 60 participants within two weeks from their baseline data collection. All patients will receive and continue their normal treatment as recommended by their primary care team. A participant may be withdrawn by the investigators, involved in major trauma or undergoes surgery, or a female participant becomes pregnant during the course of the study. Sample size was estimated using G*Power (version 3.1.5). The statistical analyses will be performed using a statistical software (IBM SPSS 22) with statistical significance set at p<0.05 for the entire analysis, unless mentioned. Descriptive statistics, interclass correlation coefficients, Bland-Altman limits of agreement plots, significance testing, correlations and regression analyses will be employed.

ELIGIBILITY:
Inclusion Criteria:

* patients with low back pain for more than three months
* aged between 18 and 65 years at baseline,
* community ambulant without walking aids,
* attending or recently attended outpatient physiotherapy treatments in the UK National Health Service (NHS) for their chronic low back pain, and
* able to read, write and understand English for completing the questionnaires

Exclusion Criteria:

* diagnosed with cancer or other self-reported specific cause [major trauma, fracture, ankylosing spondylitis, grade 3 & 4 spondylolisthesis, severe spinal canal stenosis, or lumbar intervertebral disc protrusion or extrusion, spinal deformity] for their chronic low back pain,
* underwent surgery within last one year for the lower back or are planning or scheduled for any major surgery in the coming six months,
* pregnant or experienced childbirth in the last one year,
* patients with cognitive impairment, neurological diseases, and severe vision and hearing impairments

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include community ambulant adult patients attending or recently attended outpatient physiotherapy treatment for their chronic low back pain.
Sampling Method: Non-Probability Sample
Enrollment: 270 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Change in Health Education Impact Questionnaire | baseline and 6-month follow up

SECONDARY OUTCOMES:
Duration of low back pain | baseline
Numeric Pain Intensity Scale | baseline and 6-month follow up
Roland Morris Disability Questionnaire | baseline and 6-month follow up
International Physical Activity Questionnaire (Short Form) | baseline and 6-month follow up
Tampa Scale of Kinesiophobia | baseline and 6-month follow up
Pain Catastrophising Scale | baseline and 6-month follow up
Patient Health Questionnaire 9 | baseline and 6-month follow up
Patients Global Impression of Change | 6-month follow up

CONTACTS AND LOCATIONS:
Overall Officials: Paul Hendrick, PhD, Principal Investigator — University of Nottingham
Locations (2):
- United Kingdom (2):
  - Nottingham CityCare Partnership, Nottingham, Nottinghamshire
  - Nottingham University Hospitals NHS Trust, Nottingham, Nottinghamshire

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Banerjee A, Hendrick P, Blake H. Predictors of self-management in patients with chronic low back pain: a longitudinal study. BMC Musculoskelet Disord. 2022 Dec 7;23(1):1071. doi: 10.1186/s12891-022-05933-2. PMID 36476492